CLINICAL TRIAL: NCT04261010
Title: TNF and IL23 Blocking Agents Gene Expression Ratios in the Psoriatic Arthritis Synovium
Brief Title: TNF and IL23 Blocking Agents Gene Expression Ratios in the Psoriatic Arthritis Synovium_(TIGERS) Study
Acronym: TIGERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Janssen-Cilag International NV (Industry); University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P1200_32 (TIGERS); 2017-003249-18 (EudraCT Number); FAGG/R&D/SEJ/sej (Other: FAMHP)
Record Dates: First submitted 2020-01-21; First posted 2020-02-07 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Psoriatic Arthritis
Keywords: Synovium, Biologics, Genomics
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Intervention Model Description: Randomization 1:1:1
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ustekinumab (Experimental): Group 1 (n=12): ustekinumab 45 mg (or 90 mg for patients > 100 kg) subcutaneously at baseline (W0), 4 weeks later (W4), and every 12 weeks until week 24 (i.e. W0, W4, and W16).
  Interventions: Procedure: Global/single cell gene expression profiles obtained from Synovial biopsies
- Guselkumab (Experimental): Group 2 (n=12): guselkumab 100 mg subcutaneously (regardless of the weight of the patient) at weeks 0 and 4, followed by a maintenance dose every 8 weeks through week 24 (i.e. W0, W4, W12 and W20).
  Interventions: Procedure: Global/single cell gene expression profiles obtained from Synovial biopsies
- ADALIMUMAB (Active Comparator): Group 3 (n=12): adalimumab 40 mg (regardless of the weight of the patient), subcutaneously every other week, starting from the baseline until week 24 (i.e.W0, W2, W4, W6, W8, W10, W12, W14, W16, W18, W20 and W22).
  Interventions: Procedure: Global/single cell gene expression profiles obtained from Synovial biopsies

INTERVENTIONS:
Procedure: Global/single cell gene expression profiles obtained from Synovial biopsies — Global/single cell gene expression profiles obtained from synovial biopsies before and after 24 weeks of treatment with the drug.

SUMMARY:
This study compare the genomics profiles in synovial biopsies obtained prior to, and 24 weeks after a biologic disease modifying anti-rheumatic drugs (DMARDs)(Adalimumab, Ustekinumab, Guselkumab) in patients with active psoriatic arthritis despite a treatment with a conventional synthetic DMARDs (such as methotrexate).

DETAILED DESCRIPTION:
1. STUDY SYNOPSIS 1.1 Rationale Psoriatic arthritis (PsA) is a chronic inflammatory disease, leading to impaired function, reduced quality of life, comorbidities and increased mortality. Fortunately, improved knowledge about disease mechanisms catalyzed rapid development of effective targeted therapies for this disease. PsA is a clinically heterogenous disease. Connections between clinical manifestations, disease activity, disease severity and entheseal/synovial molecular patterns are still not understood. In addition, although many treatments targeting different molecules or cytokines are now available, clinicians are still facing difficulties in the treatment choice, owing to the lack of reliable markers improving patients stratification. In the present project, we want to take advantage of our expertise in the field to compare global molecular profiles up- or down-regulated in synovitis of patients with PsA resistant to conventional synthetic disease modifying anti-rheumatic drugs (csDMARDs), before and after administration of targeted therapies, in order to identify molecular markers associated with response to therapy. This may allow us to move further towards precision medicine.

   1.2 Aim of the study We intend to evaluate global transcriptomic effects of ustekinumab (IL-12/IL-23/p40 blocker) and guselkumab (IL-23/p19 blocker) in synovial biopsies from csDMARD-resistant, biologic-naive patients with PsA, obtained prior to and 24 weeks after initiation of therapy. In parallel, synovial biopsies will be obtained before and after initiation of adalimumab (a widely used TNFα blocker) to evaluate the different molecular pathways affected by the different drugs. In order to deliver, this project will be based on the use of an Affymetrix platform (GeneChip HGU133 Plus2.0 chips). We and others amply demonstrated the power of this analytical approach in identifying synovial pathways associated with disease activity and response to therapy in the past (resulting in the development of a diagnostic and theranostic commercial kit). However, the material collected throughout the study will be a unique opportunity to carry out a more exploratory single cell RNASeq procedure on our samples, thereby potentially unravelling molecular effects of therapies in specific cell populations. Identification of the synovial effects of those treatments in psoriatic arthritis will be a step forward in understanding not only the mode of action of the drug at the site of inflammation, but also in the identification of molecular patterns associated with good response to therapy. The main advantage of our approach compared to other biomarker studies, is that we use synovial material as such, and not peripheral blood, which is a more remote location in terms of cellular targets of the drug. This project takes advantage of our strong experience in the field of molecular profiling of synovial biopsies, and evaluation of responses to biological agents. Key to the success of our translational approach is the association of reliable molecular techniques with a well-validated clinical evaluation of disease activity and response to therapy, using a panel of clinical, biological and imaging techniques.

   1.3 Study design Dual centre, 24-week open-label randomised study in subjects with clinically active peripheral PsA receiving treatment with the relevant drugs. Synovial biopsies will be obtained from patients before and after 24 weeks of treatment with the different drugs.

   1.4 Study population DMARD-resistant, biological naive patients with a diagnosis of psoriatic arthritis according to the CASPAR criteria with at least one swollen joint (either small or big joint) who are planning to receive treatment with one of the targeted drugs. In total, 36 patients will be included. Patients will be randomized 1:1:1 between: Group 1 (n=12): ustekinumab 45 mg (or 90 mg for patients > 100 kg) subcutaneously at baseline (W0), 4 weeks later (W4), and every 12 weeks until week 24 (i.e. W0, W4, and W16). Group 2 (n=12): guselkumab 100 mg subcutaneously (regardless of the weight of the patient) at weeks 0 and 4, followed by a maintenance dose every 8 weeks through week 24 (i.e. W0, W4, W12 and W20). Group 3 (n=12): adalimumab 40 mg (regardless of the weight of the patient), subcutaneously every other week, starting from the baseline until week 24 (i.e.W0, W2, W4, W6, W8, W10, W12, W14, W16, W18, W20 and W22).

   1.5 Synovial biopsy procedure Synovial biopsies will be harvested either by ultrasound guided biopsy (USGB) for small joints (wrist, MCP, PIP), or large joints (elbow, knee, ankle) or by needle-arthroscopy procedure (NAP) for large joints such as the knee.

   In the case of large joint involvement, the same joint will be biopsied at W0 and W24. Based on our experience, repeating the procedure in a large joint, even if it is not swollen, is readily achieved by NAP.

   In the case of small joint involvement, the choice of the joint to biopsy will be based on ultrasound (US) examination. An US assessment with a score of more than 2 on Grey Scale/Power Doppler (see data on US scoring below in appendices) increases the amount of gradable synovial tissue after the procedure, and the quality of the RNA extracted from the synovial tissue.

   If the small joint biopsied at W0 is not clinically affected and/or has low US Grey Scale/Power Doppler scores lower by W24, another small joint will be considered for the biopsy if clinically affected. However, At W24 the procedure will be done preferably in the same joint, in order to avoid bias or too much heterogeneity in the analyses of the data.

   A window of no more than 15 days is allowed around the baseline (W0) and W24 visit.

   1.6 Main study parameters/endpoints

   Primary endpoints:
   * identification of molecular pathways targeted by ustekinumab, guselkumab versus TNF-blockade in synovial biopsies (total and single cells) from PsA patients with active disease despite a csDMARDs, obtained prior to and 24 weeks after initiation of therapy.

   Secondary endpoints:

   - clinical response at W24, by using DAS-44 or ACR20/50/70 response criteria.

   - identification of candidate synovial markers/pathways associated with response to ustekinumab, guselkumab, and anti-TNFalpha therapy in PsA by correlating molecular signals at baseline with the clinical response observed at week 24.

   - composite analyses of the association between molecular changes induced by anti-IL23, anti-IL23/12 and anti-TNF in the synovium, and core or non-core (clinical, biological, imaging) variables informative about response to therapy.

   1.7 Clinical Assessment of disease activity Disease activity will be evaluated at screening, baseline (week 0), week 6, week 12, week 18, and week 24. Response to therapy will be evaluated at the same time using validated clinical measures of joint, enthesis and skin disease activity and global health assessment questionnaires.

   1.8 Laboratory Analyses Biochemical analysis will be performed at each visit (W0, W6, W12, W18, W24). This include C-reactive protein, liver enzymes (GOT, GPT, GGT, Alk. Phosphatase), renal function (urea, creatinin, glomerular filtration), hemogram, glycemia, lipid's profile (total cholesterol, LDL, HDL, Triglycerids).

   HLA-B27 and viral infection (hepatitis B and C, HIV) status will be checked at the screening or baseline, as well as skin PPD test or blood quantiferon-TB GOLD test.

   Blood samples (Serum, plasma, EDTA, PaxGene tubes Peripheral blood mononuclear cell (PBMC) analysis) will also be taken and or stored for further analysis 1.9 Synovial tissue analyses Affymetrix Platform (will be performed by UCL_SSS/IREC/RUMA and CUSL Site team for both sites) (at least 4 biopsy fragments/individual) RNA will be extracted from the material (at least 4 pieces) and used for hybridization of high-density oligonucleotide-spotted microarrays (Genechip U133 Plus 2.0 slides). Clustering and statistical analyses will be performed using Genespring® software in order to identify transcripts regulated by the administration of ustekinumab, guselkumab and TNF-blockade, and to identify transcripts associated with response to either of these drugs. Web-based GO and KEGG pathways mining tools will be used in order to identify potential groups of genes belonging to the same family.

   Single-cell RNA sequencing (will be performed by UZGhent Site team for both sites) (2 to 4 biopsies) If there are enough biopsies obtained, single cell analyses will be performed by UZG team. Single-cell RNA sequencing has emerged as an indispensable tool to dissect the cellular heterogeneity and decompose tissues into cell types and/or cell states, which offers enormous potential for de novo discovery. Single-cell transcriptomic atlases provide unprecedented resolution to reveal complex cellular events and deepen our understanding of biological systems.

   Histology / Immunohistochemistry (2 to 4 biopsies will be performed by CUSL Site) If there is enough tissue, part of the samples (2 biopsies) will be used for pathological examinations and standard immunohistochemistry (CD3, CD4, CD8, CD15, CD20, CD68 and CD138 immunostainings). Additional stains will be performed in order to confirm the transcriptomic results, or based on pre-established questions (Th1, Th17-specific markers).

   1.10 Imaging
   * Chest x-ray A posterior-anterior view chest x-ray will be obtained locally at screening, unless results from a chest x-ray obtained no more than 3 months prior to the screening (or baseline) according to the general recommendations related to the use of biologics.

   The chest x-ray will be reviewed by the investigator or designee to exclude patients with active TB infection.

   Investigators should follow local guidelines for monitoring patients for TB if a patient is at high risk for acquiring TB or reactivation of latent TB

   • Ultrasound: In parallel to clinical assessment, musculoskeletal ultrasound (US) will be performed at baseline (W0), W6, W12, and W24 to evaluate disease activity, with a specific focus on joints and enthesis.

   • Magnetic resonance imaging: Whole-body magnetic resonance imaging (WBMRI) evaluation will be performed at two time points, prior to initiation of therapy and 24 weeks after treatment onset, as an additional assessment tool of disease activity. Patients with any contraindications to MRI (e.g. pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments, foreign objects in the eyes, skin or body or severe claustrophobia) will not performed this procedure MRI scans will be acquired using routine scanning techniques appropriate for measurement of inflammation, bone marrow edema and erosion. The images will be analyzed locally. The readings of the scan will be performed locally.

   1.11 Study duration Study duration: 3 years

   • Screening period will start: december 2019

   • Estimated first patient inclusion (FPI): january 2020

   • Estimated last patient inclusion (LPI): january 2023

   • Estimated last patient last visit (LPLV): june 2023

   • End of Study : sept 2023
   * Publication summary: december 2023
   * Final report: october 2023

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to fulfil all of the following criteria:

1. Patient must be able to understand and communicate with the investigator and comply with the requirements of the study and must give a written, signed and dated informed consent before any study assessment is performed.
2. Male or non-pregnant, non-nursing female patients at least 18 years of age. Before randomization, a woman of childbearing potential must be on a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: eg, established use of oral, injected or implanted hormonal methods of contraception associated with inhibition of ovulation; placement of an intrauterine device (IUD) or intrauterine system (IUS); male partner sterilization (the vasectomized partner should be the sole partner for that subject); true abstinence (when this is in line with the preferred and usual lifestyle of the subject).

   A woman of childbearing potential must have a negative serum (β-human chorionic gonadotropin [β-hCG]) at baseline before randomization. A woman must agree not to donate ovocytes for the purposes of assisted reproduction during the study and for 3 months after receiving the last dose of study agent.

   Note: If the childbearing potential changes after start of the study (eg, woman who is not heterosexually active becomes active, premenarchal woman experiences menarche) that woman must begin a highly effective method of birth control, as described above.

   A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control eg, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study agent

   The method of birth control will be clearly documented in patient file.
3. Patients with active PsA according to CASPAR criteria for ≥6 months, despite ≥3 months of csDMARD therapy, and ≥4 weeks of non-steroidal anti- inflammatory drugs (NSAIDs) therapy.
4. At least 1 swollen joint at screening or baseline (despite csDMARD therapy) with ability to perform a synovial biopsy at W0.
5. Patients with newly documented latent TB are eligible provided initiation of appropriate treatment.
6. Concomitant MTX or SSZ is permitted if started ≥3 months prior to study start and at a stable dose (≤25 mg/week for MTX and ≤ 3 g/day for SSZ) for ≥4 weeks.
7. Patients on MTX must be on stable folic acid supplementation before randomization.
8. Concomitant NSAIDs and oral corticosteroids (≤10 mg prednisone/day) are permitted if stable for at least 2 weeks.
9. Allowed concomitant medications are to remain stable through week 24.
10. Patients cannot have previously received any biologic agent
11. DMARDs other than MTX or sulfasalazine (SSZ) must be interrupted. DMARDs other than MTX are not allowed within 4 weeks prior to or during trial participation. A washout period needs to be considered. (8 weeks for leflunomide).
12. At least one joint (small or large) to biopsy in order to get synovial tissue. Small joints must have an US grey-scale score > 2 on Doppler

Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for inclusion in this study.

1. Contraindications for needle-arthroscopy such as joint replacement (in the affected knee or ankle joint) or anticoagulation.
2. Use of any investigational drug and/or devices within 4 weeks of baseline, or a period of 5 half-lives of the investigational drug, whichever is longer.
3. Conditions/situations such as:

   1. Patients with conditions/concomitant diseases making them non evaluable for the primary endpoint
   2. Impossibility to meet specific protocol requirements (e.g. blood sampling)
   3. Patient is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
   4. Uncooperative or any condition that could make the patient potentially noncompliant to the study procedures
4. Any therapy by intra-articular injections (e.g. corticosteroid) within 4 weeks before baseline.
5. Any intramuscular corticosteroid injection within 2 weeks before baseline.
6. Prior treatment with a biologic agent.
7. A history of active tuberculosis (TB).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Quantitative measurement of the molecular changes in relation to the up-regulated or down-regulated genes in the synovium. | 24 weeks
  The primary endpoint of the study is not the comparative efficacy of the 3 drugs, but the comparative molecular changes they induce in the synovium.
  In a first set of analyses, the magnitude of fold-changes in (global and single cell) gene expression profiles between baseline and W24 will be analysed in each group. The higher values correspond to the high intensity in the up-regulation or down-regulation of the gene expression.

SECONDARY OUTCOMES:
Comparison between the magnitude of molecular changes (up-regulation or down-regulation of the genes) and clinical changes (improvement or worsening of the swollen joints count). | 24 weeks
  The swollen joints count (0 to 66) will be assessed. Lowered scores correspond to an improvement (remission or low disease activity), and increased value to a worsening of the clinical conditions (high disease activity). The value of the joints count will be compared to the magnitude of the up-regulation or down-regulation in the gene expression profiles.
Comparison between the magnitude of molecular changes (up-regulation or down-regulation of the genes) and imaging changes on ultrasound (US). | 24 weeks
  Synovitis (inflammation in the synovium) is scored by US in Grey-Scale (GS) (0 to 3) and Power Doppler (PD) (0 to 3). 0 correspond to lack of inflammation, and 3 to high amount of inflammation. The US changes in GS and PD will be compared to the magnitude of up-regulation or down-regulation in the gene expression profiles.
Comparison between the magnitude of molecular changes (up-regulation or down-regulation of the genes) and imaging changes on Magnetic Resonance Imaging (MRI). | 24 weeks
  MRI assessments for synovitis or bone marrow edema (water in the bone's head related to inflammation) will be binary (0 for absence of inflammation, and 1 for presence). MRI changes will be compared to the magnitude of up-regulation or down-regulation in the gene expression profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Adrien NZEUSSEU TOUKAP, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Dirk ELEWAUT, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Dirk ELEWAUT, Ghent, East Flanders
  - Adrien NZEUSSEU TOUKAP, Brussels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ritchlin CT, Colbert RA, Gladman DD. Psoriatic Arthritis. N Engl J Med. 2017 Mar 9;376(10):957-970. doi: 10.1056/NEJMra1505557. No abstract available. PMID 28273019
- [Background] Nzeusseu Toukap A, Galant C, Theate I, Maudoux AL, Lories RJ, Houssiau FA, Lauwerys BR. Identification of distinct gene expression profiles in the synovium of patients with systemic lupus erythematosus. Arthritis Rheum. 2007 May;56(5):1579-88. doi: 10.1002/art.22578. PMID 17469140
- [Background] Lauwerys BR, Hernandez-Lobato D, Gramme P, Ducreux J, Dessy A, Focant I, Ambroise J, Bearzatto B, Nzeusseu Toukap A, Van den Eynde BJ, Elewaut D, Gala JL, Durez P, Houssiau FA, Helleputte T, Dupont P. Heterogeneity of synovial molecular patterns in patients with arthritis. PLoS One. 2015 Apr 30;10(4):e0122104. doi: 10.1371/journal.pone.0122104. eCollection 2015. PMID 25927832
- [Background] De Groof A, Ducreux J, Humby F, Nzeusseu Toukap A, Badot V, Pitzalis C, Houssiau FA, Durez P, Lauwerys BR. Higher expression of TNFalpha-induced genes in the synovium of patients with early rheumatoid arthritis correlates with disease activity, and predicts absence of response to first line therapy. Arthritis Res Ther. 2016 Jan 20;18:19. doi: 10.1186/s13075-016-0919-z. PMID 26792343
- [Background] Badot V, Galant C, Nzeusseu Toukap A, Theate I, Maudoux AL, Van den Eynde BJ, Durez P, Houssiau FA, Lauwerys BR. Gene expression profiling in the synovium identifies a predictive signature of absence of response to adalimumab therapy in rheumatoid arthritis. Arthritis Res Ther. 2009;11(2):R57. doi: 10.1186/ar2678. Epub 2009 Apr 23. PMID 19389237
- [Background] Badot V, Durez P, Van den Eynde BJ, Nzeusseu-Toukap A, Houssiau FA, Lauwerys BR. Rheumatoid arthritis synovial fibroblasts produce a soluble form of the interleukin-7 receptor in response to pro-inflammatory cytokines. J Cell Mol Med. 2011 Nov;15(11):2335-42. doi: 10.1111/j.1582-4934.2010.01228.x. PMID 21129157
- [Background] Gutierrez-Roelens I, Galant C, Theate I, Lories RJ, Durez P, Nzeusseu-Toukap A, Van den Eynde B, Houssiau FA, Lauwerys BR. Rituximab treatment induces the expression of genes involved in healing processes in the rheumatoid arthritis synovium. Arthritis Rheum. 2011 May;63(5):1246-54. doi: 10.1002/art.30292. PMID 21337318
- [Background] Ducreux J, Durez P, Galant C, Nzeusseu Toukap A, Van den Eynde B, Houssiau FA, Lauwerys BR. Global molecular effects of tocilizumab therapy in rheumatoid arthritis synovium. Arthritis Rheumatol. 2014 Jan;66(1):15-23. doi: 10.1002/art.38202. PMID 24449571
- [Background] Burmester GR, Panaccione R, Gordon KB, McIlraith MJ, Lacerda AP. Adalimumab: long-term safety in 23 458 patients from global clinical trials in rheumatoid arthritis, juvenile idiopathic arthritis, ankylosing spondylitis, psoriatic arthritis, psoriasis and Crohn's disease. Ann Rheum Dis. 2013 Apr;72(4):517-24. doi: 10.1136/annrheumdis-2011-201244. Epub 2012 May 5. PMID 22562972
- [Background] McInnes IB, Mease PJ, Ritchlin CT, Rahman P, Gottlieb AB, Kirkham B, Kajekar R, Delicha EM, Pricop L, Mpofu S. Secukinumab sustains improvement in signs and symptoms of psoriatic arthritis: 2 year results from the phase 3 FUTURE 2 study. Rheumatology (Oxford). 2017 Nov 1;56(11):1993-2003. doi: 10.1093/rheumatology/kex301. PMID 28968735
- [Background] Sherlock JP, Joyce-Shaikh B, Turner SP, Chao CC, Sathe M, Grein J, Gorman DM, Bowman EP, McClanahan TK, Yearley JH, Eberl G, Buckley CD, Kastelein RA, Pierce RH, Laface DM, Cua DJ. IL-23 induces spondyloarthropathy by acting on ROR-gammat+ CD3+CD4-CD8- entheseal resident T cells. Nat Med. 2012 Jul 1;18(7):1069-76. doi: 10.1038/nm.2817. PMID 22772566
- [Background] Lories RJ, McInnes IB. Primed for inflammation: enthesis-resident T cells. Nat Med. 2012 Jul 6;18(7):1018-9. doi: 10.1038/nm.2854. No abstract available. PMID 22772553
- [Background] McInnes IB, Kavanaugh A, Gottlieb AB, Puig L, Rahman P, Ritchlin C, Brodmerkel C, Li S, Wang Y, Mendelsohn AM, Doyle MK; PSUMMIT 1 Study Group. Efficacy and safety of ustekinumab in patients with active psoriatic arthritis: 1 year results of the phase 3, multicentre, double-blind, placebo-controlled PSUMMIT 1 trial. Lancet. 2013 Aug 31;382(9894):780-9. doi: 10.1016/S0140-6736(13)60594-2. Epub 2013 Jun 13. PMID 23769296
- [Background] Kavanaugh A, Ritchlin C, Rahman P, Puig L, Gottlieb AB, Li S, Wang Y, Noonan L, Brodmerkel C, Song M, Mendelsohn AM, McInnes IB; PSUMMIT-1 and 2 Study Groups. Ustekinumab, an anti-IL-12/23 p40 monoclonal antibody, inhibits radiographic progression in patients with active psoriatic arthritis: results of an integrated analysis of radiographic data from the phase 3, multicentre, randomised, double-blind, placebo-controlled PSUMMIT-1 and PSUMMIT-2 trials. Ann Rheum Dis. 2014 Jun;73(6):1000-6. doi: 10.1136/annrheumdis-2013-204741. Epub 2014 Feb 19. PMID 24553909
- [Background] Deodhar A, Gottlieb AB, Boehncke WH, Dong B, Wang Y, Zhuang Y, Barchuk W, Xu XL, Hsia EC; CNTO1959PSA2001 Study Group. Efficacy and safety of guselkumab in patients with active psoriatic arthritis: a randomised, double-blind, placebo-controlled, phase 2 study. Lancet. 2018 Jun 2;391(10136):2213-2224. doi: 10.1016/S0140-6736(18)30952-8. Epub 2018 Jun 1. PMID 29893222
- [Background] Ritchlin C, Rahman P, Kavanaugh A, McInnes IB, Puig L, Li S, Wang Y, Shen YK, Doyle MK, Mendelsohn AM, Gottlieb AB; PSUMMIT 2 Study Group. Efficacy and safety of the anti-IL-12/23 p40 monoclonal antibody, ustekinumab, in patients with active psoriatic arthritis despite conventional non-biological and biological anti-tumour necrosis factor therapy: 6-month and 1-year results of the phase 3, multicentre, double-blind, placebo-controlled, randomised PSUMMIT 2 trial. Ann Rheum Dis. 2014 Jun;73(6):990-9. doi: 10.1136/annrheumdis-2013-204655. Epub 2014 Jan 30. PMID 24482301